CLINICAL TRIAL: NCT02593149
Title: Product Evaluation for the Effectiveness of the ClearGuard® HD End Cap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pursuit Vascular, Inc. (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0002
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): ClearGuard HD End Cap
  Interventions: Device: ClearGuard HD End Cap
- Control (No Intervention): Tego® connector with the CurosTM for Tego disinfecting port protector

INTERVENTIONS:
Device: ClearGuard HD End Cap — The ClearGuard HD end cap elutes chlorhexidine acetate into the hemodialysis hub
  Arms: Treatment

SUMMARY:
To assess blood stream infections in participants using two FDA-cleared devices: ClearGuard HD end caps compared to the Tego® connector with the CurosTM for Tego disinfecting port protector.

DETAILED DESCRIPTION:
Prospective, cluster-randomized, open-label, post market, comparative effectiveness evaluation with facilities participating for up to 13 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients dialyzing with a central venous catheter

Exclusion Criteria:

* Known allergy to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Brunelli, MD, MSCE, Principal Investigator — DaVita Clinical Research / DaVita HealthCare Partners
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brunelli SM, Van Wyck DB, Njord L, Ziebol RJ, Lynch LE, Killion DP. Cluster-Randomized Trial of Devices to Prevent Catheter-Related Bloodstream Infection. J Am Soc Nephrol. 2018 Apr;29(4):1336-1343. doi: 10.1681/ASN.2017080870. Epub 2018 Feb 22. PMID 29472415
- See also: Pursuit Vascular website — http://pursuitvascular.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline characteristic data were not collected for the participants in the "Intervention" Period. Baseline data were collected for the "Run-In" Period with the a priori intent of showing that baseline characteristics were similar in both arms. 9 patients were excluded due to heparin allergies prior to enrollment during the "Intervention" period.
Units Other Than Participants: facilities
Period: Run-In
Arm/Group | Treatment | Control
Started | 340; 20 facilities | 361; 20 facilities
Completed | 304; 20 facilities | 323; 20 facilities
Not Completed | 36; 0 facilities | 38; 0 facilities
Not completed — Didn't use CVC for at least 21 days | 36 | 38
Period: Intervention
Arm/Group | Treatment | Control
Started | 942; 20 facilities | 960; 20 facilities
Completed | 826; 20 facilities | 845; 20 facilities
Not Completed | 116; 0 facilities | 115; 0 facilities
Not completed — Didn't use CVC for at least 21 day | 116 | 115

BASELINE CHARACTERISTICS:
Population: Baseline characteristic data were not collected for the participants in the "Intervention" Period. Baseline data were collected during the "Run-In" Period with the a priori intent of demonstrating that baseline characteristics are generally balanced for the participants coming in for treatment."
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 304 | 323 | 627
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (15.6) | 62.2 (15.5) | 62.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 160 | 319
  Male | 145 | 163 | 308
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 37 | 36 | 73
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 107 | 149 | 256
  White | 133 | 122 | 255
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 13 | 37
Region of Enrollment [Number; unit: participants]
  United States | 304 | 323 | 627

OUTCOME MEASURES:

1. Primary Outcome: Positive Blood Cultures (PBC's) Per 1,000 Central Venous Catheter (CVC)-Days
Description: This was calculated by dividing the cumulative number of PBCs by cumulative time at-risk as follows.
  The National Healthcare Safety Network (NHSN) Center for Disease Control (CDC) 21-day outpatient hemodialysis patient rule is as follows: A PBC is considered a new event and counted only if it occurred 21 days or more after a previously reported PBC in the same patient; new PBC events are based on blood cultures drawn as an outpatient or within one calendar day after a hospital admission. Following a PBC additional same-type events were counted beginning 21 days following the initial event; the CVC-days were counted during this period. The CVC-days were calculated by summing the number of days each patient was at-risk of accruing a PBC. This analysis included all subjects that participated in the study that were not otherwise censored to more accurately count CVC-days.
Time Frame: Through the 13-month intervention period.
Measure: Number; unit: PBCs per 1,000 CVC-days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 826 | 845
PBCs per 1,000 CVC-days | 0.28 | 0.75

ADVERSE EVENTS:
Time Frame: 13 months
Description: The run-in data was used to determine pre-study demographics and PBC rate. No adverse event analysis was performed for this period since these patients were not enrolled in the study. This was a pragmatic post market study. There was an informed consent waiver and there were no study case report forms (CRF's). Treatment arm adverse events were monitored during the 13-month intervention period using the FDA Manufacturer and User Facility Device Experience (MAUDE) database.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/826 | 0/845
Serious Adverse Events (participants affected / at risk) | 0/826 | 0/845
Other Adverse Events (participants affected / at risk) | 0/826 | 0/845

LIMITATIONS AND CAVEATS:
This was a pragmatic post market study. There was an informed consent waiver and no CRF's. Treatment arm adverse events during the 13-month intervention period were monitored using the FDA MAUDE database and none were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No